CLINICAL TRIAL: NCT03561688
Title: Foot Orthotic for Early Stage Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionshospital Nordjylland (Other Government)
Collaborators: TrygFonden, Denmark (Industry); The Danish Rheumatism Association (Other); Aalborg University (Other); King Christian X´Hospital for Rheumatic Diseases (Other)
Responsible Party: Principal Investigator, Morten Bilde Simonsen, Principal Investigator, Regionshospital Nordjylland
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RHN_MBS_01
Record Dates: First submitted 2018-05-08; First posted 2018-06-19 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Rheumatoid Arthritis; Rheumatoid Arthritis of Foot (Disorder)
Keywords: Biomechanics; Pain; Gait; Foot orthotics; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain

STUDY DESIGN:
Intervention Model Description: The study design is a cross over study. Patients is instructed in using a placebo FO for one month and receive a custom-made FO, which they will be using for one month.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard insole (Sham Comparator): a flat insole
  Interventions: Device: Standard insole
- Foot orthotics (Experimental): Custom-made foot orthoses
  Interventions: Device: Foot orthotics

INTERVENTIONS:
Device: Foot orthotics — Insoles for shoes
  Arms: Foot orthotics
Device: Standard insole — Sham foot orthotic
  Arms: Standard insole

SUMMARY:
The overall purpose of this project is to investigate the neuro adaptations of pain and biomechanical differences between placebo and a custom-made foot orthoses for patients with RA.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is an autoimmune, chronic, progressive, systemic inflammatory disease leading to substantial pain, disability, and other morbidities. In Denmark there are 40.000 patients with RA. In RA, synovitis, effusion, eventually erosive arthritis, bone loss and weakening of the muscle and tendon apparatus are thought to cause clinically recognizable valgus heel or pes planovalgus deformity. These symptoms gradually cause irreversible joint deformities and changes in the locomotion of muscles3. Over 85% of patients with RA experience painful feet and ankles during the course of the disease. Despite medical developments, foot orthotics (FO) are still an important adjunct treatment and are often prescribed with the intention to stabilize and align the foot. This is due to a number of reasons: 1) persistent foot and ankle problems still occuring even after clinical remission is reached. 2) patients with increased disease activity may have mechanical foot impairments that need treatment in conjunction with systemic management. and 3) patients, who have not responded to or are ineligible for biologic agents, continue to have active foot impairments. However, the scientific research literature within FO treatment has lagged behind clinical practice, often leading the clinician to recommend interventions based on opinion and past experience rather than published evidence9.

Production of FO is an enormous industry. Consequently, there is a great variety of products with different materials, design, manufacturing techniques and procedures. In the literature, some FO have been shown to reduce pain however there is a considerable amount for which the studies are either inconclusive or refute the effect of FO. This might be due to differences in methodology, sparse description of the orthotics and limited information on patient's disease type and stage. However, multidisciplinary studies are still limited and it is, therefore, too early to come up with guidelines about how these interventions affect the human body mechanically from current knowledge. Previous studies have primarily focused on how foot orthotics affect pain, foot function, walking speed, forefoot plantar pressure and gait parameters, while not considering the mechanical principles on which the rationales for FO were originally based. This has led to an abundance of clinical trials that are challenging to interpret, as FO clinical outcomes and FO gait mechanics have not been studied together.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RA (EUALAR 2010) without significant damage or with small erosions but without radiological subluxation in the feet, max Larsen rheumatoid arthritis score 224.
* With clinical (medical) assessed needs for orthotics (e.g. valgus ankle, pes planus, pes planus transversus, and metatarsophalangeal instability).
* In stable disease phase (no clinically recognizable, swollen joints (but sore joints)).
* In stable treatment (no change in DMARD, NSAIDs and steroid treatment the last 4 weeks).

Exclusion Criteria:

* • Patients with RA using, or regularly used FO, or orthopedic shoes within the last 3 months.

  * Clinically significant joint disease (inflammatory or degenerative) of the knee or hip joints (according to the clinician).
  * Clinically significant back disorder (according to the clinician).
  * Patients with severe ischemic or neurological sequelae in the lower extremities.
  * BMI above 32.
  * Not suitable for a MRI scan (e.g. pacemaker, pregnancy or metal within the body).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in gait mechanics | Week 4 and 8
  Gait analysis will be performed using a 3D marker-based motion capture system from Qualisys, Sweden.
  To investigate gait mechanics, detailed patient-specific musculoskeletal (MS) computer models will be created based on clinical medical images (MRI), anthropometrics and motion capture data. The models will be created utilizing a musculoskeletal computer modeling software AnyBody Modeling System (AMS). A detailed cadaver-based model The Twente Lower Extremity Model 2.0 (TLEM 2.0) is developed for AMS to obtain patient-specific architecture, scale bones, joints, and muscles attachments relative to the patient in combination with image-based morphing techniques. These models will be used to estimate joint angles, joint torques, muscle forces and joint forces of the ankle, knee and hip joint.

SECONDARY OUTCOMES:
Change in foot pressure distribution | Week 4 and 8
  Motion capture
  A pressure insole (2-3 mm thick) system (PedarX, Novel) will be placed in the patient's shoe attached to a small computer. It is a commercial available system that can measure accurate and reliable pressure distribution for monitoring local loads between the foot and the FO.
Questionnaire - Pain - Visual analog scale | Week 0, 4 and 8
  0-10 scale from no pain to highest possible.
Insole wearing time | From week 4 to 8
  Measured by temperature sensor (Orthotimer). Orthotimer is an electronic microsensor that documents the wearing time of orthopaedic devices. It is small and flat thermometer, (9 x 1 x 4.5 mm) and will be integrated in the handed-out FO. The sensor stores time, date and temperature every 15 minutes. This information allow for accurate measurements of how often the patients uses the FO.
Pain - Pressure pain threshold | Week 0, 4 and 8
  To investigate pressure pain threshold (PPT) a handheld algometer will be used. An algometer is an instrument used to measure the pain threshold in relevant areas of the leg, foot and arm. The pain threshold is defined as the point where the pressure is experienced as pain. The pressure increases gradually with an interval until the pain is experienced and the patient presses a stop button. Each measurement is repeated 3 times in each session.
Pain mapping | Week 0, 4 and 8
  Subjects will be asked to draw their perceived pain on pain mapping drawings. Drawings will be scanned and layered and averaged though MATLAB, version 2017B (The MathWorks, Inc., Natick, Massachusetts, USA). The area of Pain will be measured using ImangeJ v.1.8.0_112 (National Institutes of Health, Madison, Wisconsin, USA).
Wearable activity monitor | From week 0 to week 8
  A commercial available accelerometer based activity monitor (Polar M200) will be lent to the participants. The device will be used to monitor the participant's activity. Participants will be instructed to use the device during the two months they are involved in the project, during the placebo period and during FO treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Morten B Simonsen, MSc, Principal Investigator — Aalborg University, Department of Health Science and Technology and Centre for Clinical Research, North Denmark Regional Hospital, Aalborg University
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - King Christian X's Hospital for Rhuematic Diseases, Gråsten
  - Department for Rheumatology, Hjørring

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Simonsen MB, Hirata RP, Naesborg-Andersen K, Leutscher PDC, Horslev-Petersen K, Woodburn J, Andersen MS. Different types of foot orthoses effect on gait mechanics in patients with rheumatoid arthritis. J Biomech. 2022 Jun;139:110496. doi: 10.1016/j.jbiomech.2021.110496. Epub 2021 Apr 30. PMID 33994179